CLINICAL TRIAL: NCT05281432
Title: Evaluation of Balance in Individuals Diagnosed With Pes Planus
Brief Title: Balance in Individuals With Pes Planus
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E-10840098-604.01.01-63688
Record Dates: First submitted 2022-03-03; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Pes Planus
Keywords: Pes Planus, Balance, Static Balance, Dynamic Balance
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pes planus individuals: The aim of this study was to evaluate the static and dynamic balance status of male individuals diagnosed with pes planus.

SUMMARY:
Pes planus, one of the most common biomechanical disorders in the lower extremities, negatively affects the daily life of the individual and their competence in activities. The aim of this study was to evaluate the static and dynamic balance status of male individuals diagnosed with pes planus.

DETAILED DESCRIPTION:
METHODS: 22 volunteer patients diagnosed with pes planus in Medipol Mega University Hospital Physical Therapy and Rehabilitation Clinic will be included in the study. This study was approved by Medipol University Non-Interventional Clinical Research Ethics Committee at the meeting numbered 10840098-604.01.01-E.63688 with decision number 1027. approved. The signatures of the participants included in the study were given with the "Informed Voluntary Consent Form". Oral and written about the research.

With the "Participant Diagnosis Form", the person's name-surname, age, gender, height, weight, body mass index, contact number, Pes Planus degree, whether he has a diagnosed disease, whether he has a past disability or whether he has had surgery will be questioned. .

In the 30-45 age group, 22 volunteers with pes planus and 24 volunteers without pes planus will be included in the study. Individuals in the pes planus group will be formed at the 2nd and 3rd levels by a single physiotherapist with clinical experience, based on the Feiss line in pes planus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, aged between 30-45 years, have not had any lower extremity injury in the last 6 months, have not had any chronic lower extremity pain, have not undergone any lower extremity surgery, and have signed an informed consent form.

Exclusion Criteria:

* Those with central nervous system and visual pathology that may affect balance, patients with vestibular pathology, deformities in the waist, hip or knee joints, amputation in the lower extremity, history of lower extremity surgery, malignancy affecting the lower extremity, those who cannot communicate, those who use assistive walking devices are obese patients were not included.

Ages: 30 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Twenty-two volunteers with pes planus and 23 volunteers without pes planus in the 30-45 age group were included in the study. The individuals constituting the pes planus group were formed by a single physiotherapist with clinical experience in pes planus, taking the Feiss line as a criterion, and individuals with pes planus at the 2nd and 3rd levels.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Tandem Posture Test; | 3 minutes
  Tandem Posture test; It is a test that evaluates the static balance in which the area in contact with the ground is narrowed. After wearing the appropriate shoelaces, it is requested that one foot touches the heel of the other net and stand for 30 seconds without support. At this time, the arms are kept close to the body. It starts with the command and the tandem position is maintained until the command stops. 30 seconds or more of the stance test is successful, 30 seconds of the test is positive, and 10 seconds or less indicates the risk of falling.
Romberg Balance Test | 3 minutes
  Romberg Balance Test; The person stands upright with his feet parallel and then closes his eyes for 20-30 seconds. The tester decides on the amount of shaking subjectively. Excessive rocking or stepping during the test indicates loss of balance. If he cannot maintain this position and loses his balance, the test is positive. The same test can be performed with one foot slightly flexed at the hip and knee.
One Leg Standing Test | 2 minutes
  One Leg Standing Test; This test serves to measure balance and static standing ability. It gives information about the risk of falling of individuals. Static balances of individuals are measured by recording the duration of standing on one leg. Eyes open first. It is tried on both legs one by one. Eyes are closed and waited for 30 seconds. 2 to 4 repetitions are allowed to record the highest performance. With the eyes closed, the longest time achieved is taken into account.
Timed Get Up and Go Test (ZKYT) | 5 minutes
  Timed Get Up and Go Test (ZKYT); The person was asked to get up from the chair he was sitting in, to walk 3 meters at a safe and normal speed, to turn, to walk back, to sit back on the chair, and the time was recorded in seconds (sec). The test is initiated with the patient's feet flat on the floor and their arms resting on the armrest of the chair. Perform three repetitions and record the best result.
Berg Balance Test | 2 minutes
  Berg Balance Test; 14 proposals and each instruction score between 0-4, 0 points when the patient cannot do the activity at all, 4 points are given when he/she completes the activity independently, The highest score is 56,0-20 points balance disorder, 21-40 points acceptable balance, 41- 56 points indicate the presence of good balance. Score <45 associated with increased risk of falling
Tinetti Balance Evaluation Scale | 5 minutes
  Tinetti Balance Evaluation Scale; Tinetti is a very important test in the evaluation of balance and gait and in the evaluation of the management of daily life alone. Tinetti scale balance score is maximum 16 points, walking score is maximum 12 points, for a total of 28 points.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sa TAN, Msc, Study Director — Istanbul Medipol University, Department of Physiotherapy and Rehabilitation
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No